CLINICAL TRIAL: NCT05308069
Title: Contact Lens Optics and Visual Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A Berntsen, OD PhD (Other)
Responsible Party: Sponsor-Investigator, David A Berntsen, OD PhD, Associate Professor, University of Houston
Organization: University of Houston (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003513
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Single vision contact lens (Other): Subjects will wear a single vision soft contact lens during the study visit
  Interventions: Device: Single vision contact lens
- Multifocal contact lens (Other): Subjects will wear a multifocal soft contact lens during the study visit
  Interventions: Device: Multifocal contact lens

INTERVENTIONS:
Device: Single vision contact lens — Subjects will wear a single vision soft contact lens only during the study visit
  Other Names: comfilcon A
  Arms: Single vision contact lens
Device: Multifocal contact lens — Subjects will wear a multifocal soft contact lens only during the study visit
  Other Names: comfilcon A
  Arms: Multifocal contact lens

SUMMARY:
This study will evaluate changes in visual performance at different pupil sizes between a single vision soft contact lens and multifocal soft contact lens, and compare refractive error measured between these two lenses with an autorefractor and an aberrometer

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand the informed consent document
* 18 to 39 years of age (inclusive)
* Best corrected visual acuity of 20/25 or better in the right eye
* Refractive error from -1.00D to -8.00D with astigmatism less than or equal to -1.00D in the right eye (corneal plane)

Exclusion Criteria:

* Any ocular or systemic conditions affecting vision, refraction, or the ability to wear a soft contact lens
* History of ocular trauma or surgery causing abnormal or distorted vision
* Current Rigid Gas Permeable (RGP) contact lens wearers
* Pregnant and/or lactating females, by self-report

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Visual performance | Through completion of study visit, an average of 3 hours
  Low contrast visual performance will be measured at different pupil sizes for each subject while wearing each of the two lenses

SECONDARY OUTCOMES:
Refractive error | Through completion of study visit, an average of 3 hours
  Refractive error will be measured with an autorefractor and an aberrometer with subjects wearing each of the two lenses

CONTACTS AND LOCATIONS:
Overall Officials: David A Berntsen, OD, PhD, Principal Investigator — University of Houston College of Optometry
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No